CLINICAL TRIAL: NCT02959619
Title: Phase 1, Dose-escalating, Open-label Study of Ensartinib, an Oral ALK Inhibitor, in Patients With ALK-positive Non-Small Cell Lung Cancer
Brief Title: Ensartinib in Non-small Cell Lung Cancer Patients With Positive ALK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-28311
Record Dates: First submitted 2016-11-06; First posted 2016-11-09 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumor; Non-Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensartinib (Experimental): Escalating dose of ensartinib was orally given once er day
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Oral ensartinib was given daily at escalating doses in a 28-day cycle
  Other Names: X-396

SUMMARY:
This study is aimed to determine the maximum tolerated dose of ensartinib, an oral ALK inhibitor in Chinese patients with ALK-positive non-small cell lung cancer

DETAILED DESCRIPTION:
The initial purpose of the study is to determine the largest amount of ensartinib that can be safely given to humans. An expansion phase will be conducted to assess the preliminary anti-tumor activity in ALK-positive non-small cell lung cancer once the recommended Phase 2 dose has been established.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor malignancy
* For the expanded cohort portion of the study, patients must have NSCLC with ALK genomic alterations positive by FISH or IHC
* Eastern Cooperative Group ECOG) Performance Status score of 0 or 1
* Adequate organ system function
* Male patients willing to use adequate contraceptive measures; female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures
* Measurable disease per RECIST
* Willingness and ability to comply with the trial and follow-up procedures
* Written informed consents are required to indicate that the patients are aware of the investigational nature of the study

Exclusion Criteria:

* Current use of anticancer therapy.
* Use of an investigational drug within 14 days or 5 half-lives (whichever is shorter) prior to the first dose of ensartinib
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days.
* Chemotherapy regimens with delayed toxicity within the last 4 weeks.
* Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Prior stem cell transplant
* Patients with a known allergy or delayed hypersensitivity reaction to drugs chemically related to ensartinib or to the active ingredient of ensartinib
* Prior use of ALK TKIs with the exception of crizotinib
* Primary CNS tumors or meningeal metastasis
* Pregnant or breastfeeding female
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of ensartinib
* Clinically significant cardiovascular disease.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* Concurrent condition evaluated by investigator would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the patient to be enrolled
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 12 months
  To characterize the preliminary pharmacokinetics of single-agent ensartinib
Area under the plasma concentration versus time curve (AUC) | 12 months
  To characterize the preliminary pharmacokinetics of single-agent ensartinib
Half-life time | 12 months
  To characterize the preliminary pharmacokinetics of single-agent ensartinib

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun yat-sen Univerisity Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma Y, Pan H, Liu Y, Zhang Y, Hong S, Huang J, Weng S, Yang Y, Fang W, Huang Y, Xiao S, Wang T, Ding L, Cui L, Zhang L, Zhao H. Ensartinib in advanced ALK-positive non-small cell lung cancer: a multicenter, open-label, two-staged, phase 1 trial. J Thorac Dis. 2022 Dec;14(12):4751-4762. doi: 10.21037/jtd-22-1606. PMID 36647478